CLINICAL TRIAL: NCT02025660
Title: Does Immune-modulation Improve the Survival in Patients With Severe Sepsis? "A Proof of the Concept Study"
Brief Title: Efficacy of Mw Vaccine in Treatment of Severe Sepsis
Acronym: MISS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IP 39
Record Dates: First submitted 2013-12-25; First posted 2014-01-01 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Severe Sepsis; Septic Shock; Immune Modulation
Keywords: Mw; Mycobacterium indicum prannii; Mycobacterium w; Severe sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mw (Experimental)
  Interventions: Drug: Mw, 0.3ml x three days sc
- Saline; 0.3 ml x three days sc (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mw, 0.3ml x three days sc
  Arms: Mw
Drug: Placebo
  Arms: Saline; 0.3 ml x three days sc

SUMMARY:
Study Hypothesis Enhancement of Th-1 response with the help of a poly TLR agonist (Mw) is likely to increase survival in patients with severe sepsis.

Objectives To study whether immunomodulation with Mycobacterium Mw helps in improving survival and the recovery of organ function in patients with severe sepsis. This will be assessed with the help of the following

* Mortality in the two arms
* Daily SOFA scores
* Ventilator free days
* Time-to-vasopressor withdrawal
* ICU length of stay
* Hospital length of stay METHODS This will be a proof of the concept study to assess the effect of Mycobacterium w in combination with standard therapy versus standard therapy alone on the inflammatory profile in sepsis due to gram negative infection. A total of 25 patients will be enrolled in each group. The patients will be randomized in balance to receive either test drug or its placebo along with the standard of care

DETAILED DESCRIPTION:
This will be a proof of the concept study to assess the effect of Mycobacterium w in combination with standard therapy versus standard therapy alone on the inflammatory profile in sepsis due to gram negative infection. The study will be conducted in the respiratory intensive care unit at PGIMER, Chandigarh, over a period of 1 year. A total of 25 patients will be enrolled in each group. The patients will be randomized in balance to receive either test drug or its placebo along with the standard of care

In addition to the standard therapy for sepsis, patients randomized to test arm will receive single daily dose of 0.3 ml of Mw intra-dermal for 3 consecutive days while patients randomized to control arm will receive single daily dose of 0.3 ml of Mw-placebo intra-dermal for 3 consecutive days.

Study Duration Study duration for each patient will be 28 days. Follow up period is included in the study duration of 28 days

Study Outlines and Timing of Visits Eligible patients will be enrolled after due consent and randomized to one of the treatment arms. The enrolled patients will be monitored for any adverse events (AEs) or serious adverse events (SAEs) throughout the study period. All patients will continue to receive standard therapy till considered requisite

ELIGIBILITY:
Inclusion Criteria:

-

All consecutive patients admitted in respiratory intensive care unit of our Institute with severe sepsis or septic shock fulfilling the following criteria will be included in the study after taking the informed consent:

1. Any patient of severe sepsis or septic shock as defined below:

   • Systemic Inflammatory Response Syndrome (SIRS): Two or more of the following conditions: temperature >38.5°C or <36.0°C; heart rate of >90 beats/min; respiratory rate of >20 breaths/min or PaCO2 of <32 mm Hg; and WBC count of >12,000 cells/mL or <4000 cells/mL, or >10 percent immature (band) forms

   • Sepsis: SIRS in response to presumed or documented infection (culture or Gram stain of blood, sputum, urine, or normally sterile body fluid positive for pathogenic microorganism; or focus of infection identified by visual inspection, e.g., ruptured bowel with free air or bowel contents found in abdomen at surgery, wound with purulent discharge, consolidation on chest radiograph).

   • Severe sepsis: Sepsis and at least one of the following signs of organ hypoperfusion or organ dysfunction: areas of mottled skin; capillary refilling of 3 s; urinary output of <0.5 mL/kg for at least 1 h or renal replacement therapy; lactate >2 mmol/L; abrupt change in mental status or abnormal EEG findings; platelet count of <100,000 cells/mL or disseminated intravascular coagulation; acute lung injury/ARDS; and cardiac dysfunction (echocardiography)

   • Septic shock: Severe sepsis and one of the following conditions: Systemic mean BP of <60 mm Hg (<80 mm Hg if previous hypertension) after 40 to 60 mL/kg saline solution, or PCWP between 12 and 20 mm Hg; and Need for dopamine of >5 mcg/kg/min, or norepinephrine or epinephrine of <0.25 mcg/kg/min to maintain mean BP at >60 mm Hg (80 mm Hg if previous hypertension)

   • Refractory septic shock: Need for dopamine at >15 mcg/kg/min, or nor-epinephrine or epinephrine at >0.25 mcg/kg/min to maintain mean BP at >60 mm Hg (80 mm Hg if previous hypertension)
2. AND having at least one of the following:

   * Source of Gram negative sepsis presumed to be originating from these sources (gastrointestinal, hepatobiliary, genitourinary tract, pulmonary, neurological) or
   * Documented by typical clinical signs and symptoms and confirmed by blood culture and/or histology or
   * Documented by typical clinical signs and symptoms and confirmed by CSF culture/tissue culture and/or histology or
   * Positive culture or histology confirmation or any other investigation deemed necessary must be obtained at the time of enrolment and prior to the first dose of study medication
3. Patients and/or legally authorized representative(s), if applicable, have been fully informed and have given written informed consent. A patient unable to write and /or read but who fully understands the oral information given by the investigator (or nominated representative) has given oral informed consent witnessed in writing by an independent person.
4. Patients of either gender in the age range of 18-65 years
5. Female patients of child bearing potential must have a negative pregnancy test within 14 days prior to first dose of study medication. They must avoid becoming pregnant while receiving study medication by maintaining adequate birth control practice
6. Patients must have sufficient venous access to permit administration of medication and monitoring of safety variables.

Exclusion Criteria:

* 1. Blood culture is positive for Gram-positive organism. 2. Patient is pregnant or nursing. 3. Patients whose sole diagnosis is fungal sepsis. 4. Patients with history of allergy, hypersensitivity, or any serious reaction to study medication.

  5. Patient previously enrolled into this study. 6. Patient participating or having participated in a clinical trial with another investigational drug within the last 28 days except for investigational drugs against cancer, leukaemia or HIV.

  7. Patients with a concomitant medical condition, whose participation may create an unacceptable additional risk.

  8. Patients with a life expectancy judged to be less than five days from the basic disease other than sepsis.

  9. History of cardiopulmonary resuscitation for the current episode of sepsis 10. Patients not willing to participate or not likely to complete the trial as per judgement of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mortality | upto 4 weeks

SECONDARY OUTCOMES:
Hospital length of stay | upto 4 weeks

OTHER OUTCOMES:
ICU length of stay | upto 4 weeks
Daily SOFA score | upto 4 weeks
Vasopressor free days | upto 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inderpaul si Sehgal, Principal Investigator — PIMER, Chandigarh
Locations (1):
- PIMER, Chandigarh, Chandigarh, India